CLINICAL TRIAL: NCT04751292
Title: HIGH Altitude CArdiovascular REsearch Latin America Population Study
Acronym: HIGHCARE-LAPS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: 09A921
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Cardiovascular Risk Factor; Altitude Hypoxia; Altitude Sickness; Erythrocytosis; Sleep
Keywords: ambulatory blood pressure monitoring; echocardiography
MeSH Terms: conditions — Hypertension; Altitude Sickness; Polycythemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lowlanders: People living at low (<1500 m) altitude
- Highlanders: People living at high (>2500 m) altitude
  Interventions: Other: Exposure to high altitude

INTERVENTIONS:
Other: Exposure to high altitude — permanence at high (>2500 m) altitude; permanence is defined as being born and living at high altitude with the total time spent at lower altitudes not exceeding 2 years in the past 10 years
  Groups: Highlanders

SUMMARY:
High blood pressure (BP) is one of the principal cardiovascular risk factors. While BP levels and hypertension prevalence are well characterized in many populations, information on BP and on cardiovascular risk profile in high altitude inhabitants is limited and frequently contradictory, especially in the large highland populations of South America. The information on the effects of permanent high altitude exposure on cardiovascular variables including BP may be relevant in the light of the known BP-increasing effect of acute exposure to high altitude hypoxia. This information may have practical implications for millions of people living at elevated altitudes in Asia, South America and Africa.

The inconclusive epidemiological evidence on BP and cardiovascular risk in high altitude dwellers may be the result of several factors, among them: 1) confounding by genetic and socio-economic factors; 2) imperfect methods of BP evaluation, in particular lack of data on ambulatory and home BP (both methods considered superior to conventional clinic BP in the assessment of exposure to high BP).

On this background, the general aim of the study is to compare blood pressure levels and cardiovascular risk profile among population-based samples of subjects residing in Peruvian communities living at different altitudes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) male and female subjects;
* Highlanders: permanence at high (>2500 m) altitude;
* Lowlanders: permanence at low (<1500 m) altitude;
* Written informed consent to participate in the study

Exclusion Criteria:

* Lowlanders who over 3 months preceding inclusion in the study spent considerable (> 7 consecutive days) amount of time at altitudes above 1500 m;
* Highlanders who over 3 months preceding inclusion in the study spent considerable (>7 consecutive days) amount of time at altitudes below 2500 m;
* Subjects cognitively incapable of providing informed consent or responding to a questionnaire
* Physical disability that would prevent study assessments from being performed
* Active pulmonary tuberculosis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited by random sampling from the general population residing permanently in urban areas at:
  1. Sea level (lowlanders): <500m altitude (the city of Lima and surroundings, population 7.605.742)
  2. High altitude (highlanders):
     * 2500-3500 m (Cajamarca, 2,720 m, population 283.767; Cuzco, 3,399 m, pop. 420.137; Huancayo, 3.287m, pop. 501.384)
     * 3500-4000 m Juliaca, 3,824 m, pop. 216.716,
     * >4000 m (Ananea, 4.616m, pop. 20.572; La Rinconada 5.100m, pop. 50.000; Cerro de Pasco, 4.300-4.700 m, pop. 70.000)
Sampling Method: Probability Sample
Enrollment: 937 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in 24 h ambulatory systolic BP between lowlanders and highlanders. | baseline

SECONDARY OUTCOMES:
Differences in 24 h DBP, daytime and night-time systolic and diastolic BP between lowlanders and highlanders | baseline
Difference in conventional systolic and diastolic BP between lowlanders and highlanders | baseline
Difference in home systolic and diastolic BP between lowlanders and highlanders | baseline
Difference in sleep quality between lowlanders and highlanders | baseline
  Pittsburgh questionnaire (score)
Difference in sleep duration between lowlanders and highlanders | baseline
  self reported sleep duration (hours)
Difference in estimated cardiovascular risk | baseline
Difference between lowlanders and highlanders in hypertension prevalence | baseline
Difference in a number of BP variables between highlanders living at three high altitude levels | baseline

OTHER OUTCOMES:
Differences between lowlanders and highlanders and among highlanders living at different high altitude levels in Left Ventricular Mass assessed by echocardiography | baseline
  echocardiography, ASE convention
Differences between lowlanders and highlanders and among highlanders living at different high altitude levels in nocturnal oxygen saturation | baseline
  Cardiorespiratory sleep monitoring
Differences between lowlanders and highlanders and among highlanders living at different high altitude levels in Apnea Hypopnea Index during sleep | baseline
  Cardiorespiratory sleep monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano; Grzegorz Bilo, PhD, Study Director — Istituto Auxologico Italiano; Francisco Villafuerte, PhD, Study Director — Universidad Peruviana Cayetano Heredia
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
The data will be placed in a public repository and available upon reasonable request after study completion

REFERENCES:
- [Background] Bilo G, Acone L, Anza-Ramirez C, Macarlupu JL, Soranna D, Zambon A, Vizcardo-Galindo G, Pengo MF, Villafuerte FC, Parati G; HIGHCARE-ANDES Highlanders Study Investigators. Office and Ambulatory Arterial Hypertension in Highlanders: HIGHCARE-ANDES Highlanders Study. Hypertension. 2020 Dec;76(6):1962-1970. doi: 10.1161/HYPERTENSIONAHA.120.16010. Epub 2020 Nov 11. PMID 33175629
- [Background] Torlasco C, Bilo G, Giuliano A, Soranna D, Ravaro S, Oliverio G, Faini A, Zambon A, Lombardi C, Parati G. Effects of acute exposure to moderate altitude on blood pressure and sleep breathing patterns. Int J Cardiol. 2020 Feb 15;301:173-179. doi: 10.1016/j.ijcard.2019.09.034. Epub 2019 Oct 30. PMID 31780104
- [Background] Bilo G, Caravita S, Torlasco C, Parati G. Blood pressure at high altitude: physiology and clinical implications. Kardiol Pol. 2019 Jun 25;77(6):596-603. doi: 10.33963/KP.14832. Epub 2019 May 17. PMID 31099758
- [Background] Hainsworth R, Drinkhill MJ. Cardiovascular adjustments for life at high altitude. Respir Physiol Neurobiol. 2007 Sep 30;158(2-3):204-11. doi: 10.1016/j.resp.2007.05.006. Epub 2007 May 18. PMID 17597013
- [Background] Parati G, Agostoni P, Basnyat B, Bilo G, Brugger H, Coca A, Festi L, Giardini G, Lironcurti A, Luks AM, Maggiorini M, Modesti PA, Swenson ER, Williams B, Bartsch P, Torlasco C. Clinical recommendations for high altitude exposure of individuals with pre-existing cardiovascular conditions: A joint statement by the European Society of Cardiology, the Council on Hypertension of the European Society of Cardiology, the European Society of Hypertension, the International Society of Mountain Medicine, the Italian Society of Hypertension and the Italian Society of Mountain Medicine. Eur Heart J. 2018 May 1;39(17):1546-1554. doi: 10.1093/eurheartj/ehx720. PMID 29340578
- [Background] Duplain H, Vollenweider L, Delabays A, Nicod P, Bartsch P, Scherrer U. Augmented sympathetic activation during short-term hypoxia and high-altitude exposure in subjects susceptible to high-altitude pulmonary edema. Circulation. 1999 Apr 6;99(13):1713-8. doi: 10.1161/01.cir.99.13.1713. PMID 10190881
- [Background] Hansen J, Sander M. Sympathetic neural overactivity in healthy humans after prolonged exposure to hypobaric hypoxia. J Physiol. 2003 Feb 1;546(Pt 3):921-9. doi: 10.1113/jphysiol.2002.031765. PMID 12563015
- [Background] Bartsch P, Gibbs JS. Effect of altitude on the heart and the lungs. Circulation. 2007 Nov 6;116(19):2191-202. doi: 10.1161/CIRCULATIONAHA.106.650796. No abstract available. PMID 17984389
- [Background] Higgins JP, Tuttle T, Higgins JA. Altitude and the heart: is going high safe for your cardiac patient? Am Heart J. 2010 Jan;159(1):25-32. doi: 10.1016/j.ahj.2009.10.028. PMID 20102863
- [Background] Bilo G, Caldara G, Styczkiewicz K, Revera M, Lombardi C, Giglio A, Zambon A, Corrao G, Faini A, Valentini M, Mancia G, Parati G. Effects of selective and nonselective beta-blockade on 24-h ambulatory blood pressure under hypobaric hypoxia at altitude. J Hypertens. 2011 Feb;29(2):380-7. doi: 10.1097/HJH.0b013e3283409014. PMID 21045724
- [Background] Parati G, Bilo G, Faini A, Bilo B, Revera M, Giuliano A, Lombardi C, Caldara G, Gregorini F, Styczkiewicz K, Zambon A, Piperno A, Modesti PA, Agostoni P, Mancia G. Changes in 24 h ambulatory blood pressure and effects of angiotensin II receptor blockade during acute and prolonged high-altitude exposure: a randomized clinical trial. Eur Heart J. 2014 Nov 21;35(44):3113-22. doi: 10.1093/eurheartj/ehu275. Epub 2014 Aug 26. PMID 25161182
- [Background] Bilo G, Villafuerte FC, Faini A, Anza-Ramirez C, Revera M, Giuliano A, Caravita S, Gregorini F, Lombardi C, Salvioni E, Macarlupu JL, Ossoli D, Landaveri L, Lang M, Agostoni P, Sosa JM, Mancia G, Parati G. Ambulatory blood pressure in untreated and treated hypertensive patients at high altitude: the High Altitude Cardiovascular Research-Andes study. Hypertension. 2015 Jun;65(6):1266-72. doi: 10.1161/HYPERTENSIONAHA.114.05003. Epub 2015 Apr 20. PMID 25895588
- [Background] Savla JJ, Levine BD, Sadek HA. The Effect of Hypoxia on Cardiovascular Disease: Friend or Foe? High Alt Med Biol. 2018 Jun;19(2):124-130. doi: 10.1089/ham.2018.0044. PMID 29939783
- [Background] Aryal N, Weatherall M, Bhatta YK, Mann S. Blood Pressure and Hypertension in Adults Permanently Living at High Altitude: A Systematic Review and Meta-Analysis. High Alt Med Biol. 2016 Sep;17(3):185-193. doi: 10.1089/ham.2015.0118. Epub 2016 Aug 30. PMID 27575245
- [Background] Beall CM. Andean, Tibetan, and Ethiopian patterns of adaptation to high-altitude hypoxia. Integr Comp Biol. 2006 Feb;46(1):18-24. doi: 10.1093/icb/icj004. Epub 2006 Jan 6. PMID 21672719
- [Background] Bernabe-Ortiz A, Carrillo-Larco RM, Gilman RH, Checkley W, Smeeth L, Miranda JJ; CRONICAS Cohort Study Group. Impact of urbanisation and altitude on the incidence of, and risk factors for, hypertension. Heart. 2017 Jun;103(11):827-833. doi: 10.1136/heartjnl-2016-310347. Epub 2017 Jan 23. PMID 28115473
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] O'Brien E, Parati G, Stergiou G, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring. European Society of Hypertension position paper on ambulatory blood pressure monitoring. J Hypertens. 2013 Sep;31(9):1731-68. doi: 10.1097/HJH.0b013e328363e964. PMID 24029863
- [Background] Corante N, Anza-Ramirez C, Figueroa-Mujica R, Macarlupu JL, Vizcardo-Galindo G, Bilo G, Parati G, Gamboa JL, Leon-Velarde F, Villafuerte FC. Excessive Erythrocytosis and Cardiovascular Risk in Andean Highlanders. High Alt Med Biol. 2018 Sep;19(3):221-231. doi: 10.1089/ham.2017.0123. Epub 2018 May 21. PMID 29782186